CLINICAL TRIAL: NCT07344831
Title: Impact of Fatty Stimuli on Cerebral Activity in Anorexia Nervosa: a Multi-sensory Approach
Acronym: ANOVERSION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24CH172; ANSM (Other: 2024-A02435-42)
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa,; MRI; Lipid aversion
MeSH Terms: conditions — Anorexia Nervosa | interventions — Smell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anorexia Nervosa patient group (Experimental): 30 patients with anorexia nervosa
  Interventions: Other: MRI examination; Other: Smell and taste capacity testings
- Normal Weight Control group (Active Comparator): 30 control subjects of normal weight
  Interventions: Other: MRI examination; Other: Smell and taste capacity testings
- Low Weight Control group (Active Comparator): 30 control subjects with a similar weight to AN patients (the constitutional thinness group)
  Interventions: Other: MRI examination; Other: Smell and taste capacity testings

INTERVENTIONS:
Other: MRI examination — One hour MRI examination
Other: Smell and taste capacity testings — one hour sensory testings

SUMMARY:
Lipid restriction is significant in anorexia nervosa and limits therapeutic management. The multisensory perception of fat is altered, creating an aversion to lipids. The investigators aim to characterize the impact of sensory stimulation (smells or images) associated with specific tastes using neuropsychological assessments and functional MRI. Some volatile aromas can enhance the perception of the associated taste. The investigators hypothesize that such associations are altered in anorexia nervosa for fatty foods but may be preserved for sweet tastes, and that this alteration contributes to the maintenance of the disease. The interdependence of different sensory perceptions of lipids could play a major role in the therapeutic approach, aiding in the deconditioning of this aversion and the restoration of positive food sensory associations.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated or entitled to a social security scheme
* Person having received informed information on the study and having co-signed, with the investigator, a consent to participate in the study
* female person
* Person affiliated or entitled to a social security scheme
* Over 18 years'old
* Knowing how to read and write French
* Patient diagnosed with anorexia nervosa according to DSM-5 criteria for at least 5 years (HAS criteria). Failure of prior outpatient or/and hospitalization care over the last 12 months: stable or falling low BMI, unmodified food restriction, continued fear of weight gain, disturbances in the perception of body image
* BMI < 18.5 kg/m² for volunteers in a state of constitutional thinness. The absence of eating disorder and the absence of restriction to DEBQ questionnaires. Fertility preserved.
* For volunteers of normal weight: 18.5 kg/m² < BMI < 25 kg/m²

Exclusion Criteria:

* Pregnant women, parturient, nursing mothers;
* Persons deprived of their liberty, hospitalized without consent, hospitalized for purposes other than research;
* Minors
* Refusal of the study by the participant
* Person incapable of giving informed consent
* Artificial nutrition
* Associated organic damage favoring undernutrition: other chronic diseases (digestive, infectious, endocrine, pulmonary, cardiac, neurological), neoplasms, etc.
* Abuse of psychoactive substances except tobacco
* Characterized depressive episode, psychosis
* Score less than 14 on the Edinburgh laterality questionnaire.
* Contraindications to MRI or allergy to one of the components of the olfactory and taste tests
* Smokers
* Smell or taste alterations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Brain activity measured by functional MRI | Day 1
  Estimation of the "fatty vs. neutral" contrast when all three senses are used, comparing AN patients to the normal-weight control group (NC group) in each voxel of the brain volume (whole-brain analysis) and in the orbitofrontal cortex (ROI analysis).

SECONDARY OUTCOMES:
Brain activity measured by functional MRI | Day 1
  Estimation of the "fatty vs. neutral" contrast when all three senses are used, comparing AN patients to the control group with a similar BMI (CT group) in each voxel of the brain volume (whole-brain analysis) and in the orbitofrontal cortex (ROI analysis).
Brain activity measured by functional MRI | Day 1
  BOLD signal variations between the groups (AN, NC, and CT) for the "sweet vs. neutral" contrast.
Brain activity measured by functional MRI | Day 1
  BOLD signal variations for single vs. three senses simultaneously for each group and between groups for the "fatty vs. neutral" and "sweet vs. neutral" contrasts.
BMI | DAY 1.
  Body Mass Index
Olfactory and gustatory abilities | Day 1
  MediSens tests of olfactory and gustatory abilities
3DT1 morphological MRI | Day 1
  Brain morphometric measures and voxel-based morphometry.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No